CLINICAL TRIAL: NCT01310023
Title: Surveillance Monitoring for ART Toxicities Study in HIV Uninfected Children Born to HIV Infected Women
Acronym: SMARTT
Status: Completed | Type: Observational
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute on Drug Abuse (NIDA) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); National Institute of Mental Health (NIMH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Tulane University School of Medicine (Other); National Institute of Dental and Craniofacial Research (NIDCR) (NIH); NIH Office of AIDS Research (OAR) (NIH)
Responsible Party: Principal Investigator, Paige Williams, Senior Lecturer on Biostatistics, Harvard School of Public Health (HSPH)
Other Study IDs: 1P01HD103133 - PH100; PH100 (Other: PHACS Protocol Number); 1P01HD103133 (NIH); NCT00647803 (obsolete NCT alias)
Record Dates: First submitted 2011-03-04; First posted 2011-03-07 (Estimated); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Antiretroviral Toxicity
Keywords: Conditions and diagnoses potentially related to perinatal exposure to antiretroviral medications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, cell pellets, meconium, saliva, hair
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Static Cohort- closed to enrollment and follow-up: HIV-uninfected children < 12 years of age at the time of enrollment, born of HIV-infected mothers
- Dynamic Cohort: HIV-uninfected children born of HIV-infected mothers enrolled from prior to birth through ≤ 72 hours of age
- Reference Cohort- closed to enrollment and follow-up: HIV-uninfected children born to a mother HIV uninfected at the time of the child's birth enrolled at 1, 3, 5, or 9 years of age(± 3 months) at the time of the study visit
- Young Adult Cohort- closed to enrollment and follow-up: Former Dynamic and Static Cohort participants ≥ 18 years of age.

SUMMARY:
SMARTT will estimate the incidence of conditions and diagnoses potentially related to in utero exposure to antiretroviral therapy and/or exposure in the first two months of life among children born of HIV-infected mothers.

DETAILED DESCRIPTION:
Many antiretroviral therapy (ART) medications given to a pregnant woman cross the placenta and can be detected in the amniotic fluid and cord blood resulting in substantial fetal exposure. Therefore, there is concern about toxicity of the drugs in the fetus and infant. It is noteworthy that none of the currently approved ART medications for the prevention of maternal to fetal transmission of HIV are in Food and Drug Administration (FDA) Pregnancy Category A (no fetal risk ascertained in adequately controlled human studies). Thus, there is continued need to examine the toxicity of ART in HIV transmission prevention for the short-term toxicity of newer agents and combinations as well as the unanswered questions of longer term toxicity and subtle adverse effects.

The study will use a registry approach to conduct active surveillance among children < 12 years of age at enrollment. Occurrences of abnormalities from ART exposure in utero and/or in the first two months of life will be sought in multiple domains, including metabolic, growth, cardiac, neurologic, neurodevelopmental, behavior, language, and hearing. Clinical and laboratory data will be examined for abnormalities through a hierarchy of evaluations: adverse events (AE) will be identified → selected AEs will trigger predefined additional evaluations → significant observations will be defined as cases → a pattern of significant study-wide cases will be defined as signals. The incidence of these events of interest will be monitored over time and by ART regimen, and compared with historical data that may be suggestive of a signal. Some signals may be testable using existing and/or previously collected data, while other signals may indicate the need for additional hypothesis-driven studies outside of SMARTT.

The objectives of SMARTT are:

1. To estimate the occurrence of potential ART-related toxicities through an ongoing surveillance system among HIV-uninfected children born to mothers with HIV infection with and without exposure to ART in utero and/or in the first two months of life and compare the occurrences of these outcomes with other sources of data as well as by ART exposures; and
2. To actively encourage hypothesis-driven studies to confirm that the signals are due to ART exposure in utero and/or in the first two months of life. Note that the full design and execution of these studies may be beyond the scope of the SMARTT study but will be facilitated by SMARTT.

The specific aims of SMARTT are:

1. To create a Static Surveillance Cohort to extend domain-specific data collection in children either 1) previously enrolled in any of the approved studies for enrollment into SMARTT; 2) previously enrolled in another pediatric HIV/AIDS cohort study with SMARTT Protocol Chair approval, or 3) not previously enrolled in an approved study but with equivalent data available in the medical record;
2. To create a Dynamic Surveillance Cohort to examine domain-specific data of children newly exposed to ART in utero and/or in the first two months of life;
3. To create a Young Adult Cohort to study long-term outcomes in SMARTT participants formerly enrolled in the Static and Dynamic cohorts.
4. To identify a set of "triggers" for each domain that define a "signal" of possible ART toxicity and compare the occurrence of these signals with previously collected data and by ART exposure; and
5. To encourage and facilitate the development of hypothesis-driven studies to evaluate whether a "signal" is the result of ART exposure in utero and/or in the first two months of life.

ELIGIBILITY:
Inclusion Criteria:

Dynamic Cohort:

* HIV-exposed living fetus greater than or equal to 23 weeks gestation or a live infant born after 22 weeks gestation. Infants exposed and unexposed to ART will be enrolled.
* Any infant born of an HIV-infected mother may be enrolled pending determination of the infant's HIV infection status. However, infants found to be HIV-positive will be discontinued from the study and will be referred for care outside this study. HIV infection status will be determined using the Diagnosis of Lack of Infection in HIV-Exposed Children.
* ART exposure data by trimester of pregnancy must be available if ART exposed.
* Entry prior to birth through < 72 hours of age.
* Willingness of parent/legal guardian to provide written permission for child to participate in study.
* Willingness of biological mother to enroll at initial enrollment of her child.

Exclusion Criteria:

Dynamic Cohort:

None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Children aged 0 - < 12 years born of HIV-infected mothers recruited from a clinical setting.
Sampling Method: Non-Probability Sample
Enrollment: 5169 (Actual)
Dates: Start 2007-03; Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Neurologic abnormalities | Annually birth through age 5; semiannual thereafter, assessments vary based on age of child.
  Assessed via head circumference measurement and medical record review for documented clinical diagnoses of seizures, microcephaly, or other neurologic diagnosis.
Neurodevelopmental abnormalities | 1, 3, 5, 9, and 13 years of age, assessments vary based on age of child.
  Assessed via the following neurodevelopmental tests: Bayley Screener, Bayley III, WPPSI-III, BASC-2, WASI, WISC-IV, BRIEF, WIAT II.
Abnormal growth and metabolic function | Annually birth through age 5; semiannual thereafter, assessments vary based on age of child.
  Assessed through the measurement of height, weight, tricep skinfold thickness, mid-upperarm circumference measurements, insulin and glucose, and fasting lipids.
Cardiac abnormalities | Ages 3-5.
  Assessed through the administration of echocardiograms and serum biomarkers (ProBNP).
Hearing dysfunction | At age 5 and for children of all ages meeting a hearing/language trigger.
  Assessed via audiologic evaluation conducted by an audiologist.
Language dysfunction | 1, 2, 3, 5, and 9 years of age, assessments vary based on age.
  Assessed via the following language tests: MCDI, Ages and Stages Communication Scale, PPVT IV, Goldman Fristoe 2, Rice Wexler, TELD-3, TOLD-3, Woodcock, CELF IV.
Drug Use and Sexual Activity | 11, 13, 15, and 17 years of age.
  The assessment of sexual behavior and substance use will be conducted using an Audio Computer Assisted Survey Instrument (ACASI). ACASI uses computer and voice recordings so that the participant hears (through headphones) and sees (on the screen) each question and response list. The use of ACASI is proven to minimize response bias due to the presence of an interviewer.
Abnormal organ function | Birth and age one, semiannual thereafter.
  Assessed through the measurement of lipase, CPK, ALT, creatinine, glucose, LDH, BUN, WBC, PMN, lymphocytes, platelets, or hemoglobin ( ≥ Grade 3 adverse event).
Death due to unknown medical condition | Annual.
  Assessed through autopsy review.

SECONDARY OUTCOMES:
Maternal substance use during pregnancy | Entry visit.
  Obtained via interview, toxicology report, and meconium testing.

CONTACTS AND LOCATIONS:
Overall Officials: Paige L Williams, Principal Investigator — Harvard School of Public Health (HSPH); Ellen Chadwick, M.D., Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (22):
- United States (20):
  - University of Alabama, Birmingham, Alabama
  - University of California San Diego, La Jolla, California
  - University of Southern California, Los Angeles, California
  - University of Colorado Denver Health Sciences Center, Aurora, Colorado
  - Children's Diagnostic & Treatment Center, Fort Lauderdale, Florida
  - University of Florida Health Science Center, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - University of Illinois, Chicago, Chicago, Illinois
  - Ann and Robert H. Lurie Children's Hospital, Chicago, Illinois
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Rutgers - New Jersey Medical School, Newark, New Jersey
  - SUNY Downstate Medical Center, Brooklyn, New York
  - New York University School of Medicine, New York, New York
  - SUNY Stony Brook, Stony Brook, New York
  - Bronx Lebanon Hospital Center, The Bronx, New York
  - Jacobi Medical Center, The Bronx, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Baylor College of Medicine, Houston, Texas
- Puerto Rico (2):
  - University of Puerto Rico Medical Center, San Juan, PR
  - San Juan Research Hospital, San Juan

REFERENCES:
- [Background] Fulcher IR, Tchetgen Tchetgen EJ, Williams PL. Mediation Analysis for Censored Survival Data Under an Accelerated Failure Time Model. Epidemiology. 2017 Sep;28(5):660-666. doi: 10.1097/EDE.0000000000000687. PMID 28574921
- [Background] Correia K, Williams PL. Estimating the Relative Excess Risk Due to Interaction in Clustered-Data Settings. Am J Epidemiol. 2018 Nov 1;187(11):2470-2480. doi: 10.1093/aje/kwy154. PMID 30060004
- [Background] Correia K, Williams PL. A hierarchical modeling approach for assessing the safety of exposure to complex antiretroviral drug regimens during pregnancy. Stat Methods Med Res. 2019 Feb;28(2):599-612. doi: 10.1177/0962280217732597. Epub 2017 Oct 3. PMID 28969502
- [Background] Zash RM, Williams PL, Sibiude J, Lyall H, Kakkar F. Surveillance monitoring for safety of in utero antiretroviral therapy exposures: current strategies and challenges. Expert Opin Drug Saf. 2016 Nov;15(11):1501-1513. doi: 10.1080/14740338.2016.1226281. Epub 2016 Sep 6. PMID 27552003
- [Background] Bather JR, Horton NJ, Coull BA, Williams PL. The impact of correlated exposures and missing data on multiple informant models used to identify critical exposure windows. Stat Med. 2023 Apr 15;42(8):1171-1187. doi: 10.1002/sim.9664. Epub 2023 Jan 16. PMID 36647625
- [Result] Tassiopoulos K, Read JS, Brogly S, Rich K, Lester B, Spector SA, Yogev R, Seage GR 3rd. Substance use in HIV-Infected women during pregnancy: self-report versus meconium analysis. AIDS Behav. 2010 Dec;14(6):1269-78. doi: 10.1007/s10461-010-9705-0. PMID 20532607
- [Result] Griner R, Williams PL, Read JS, Seage GR 3rd, Crain M, Yogev R, Hazra R, Rich K; Pediatric HIV/AIDS Cohort Study. In utero and postnatal exposure to antiretrovirals among HIV-exposed but uninfected children in the United States. AIDS Patient Care STDS. 2011 Jul;25(7):385-94. doi: 10.1089/apc.2011.0068. Epub 2011 Jun 10. PMID 21992592
- [Result] Crain MJ, Williams PL, Griner R, Tassiopoulos K, Read JS, Mofenson LM, Rich KC; Pediatric HIVAIDS Cohort Study. Point-of-care capillary blood lactate measurements in human immunodeficiency virus-uninfected children with in utero exposure to human immunodeficiency virus and antiretroviral medications. Pediatr Infect Dis J. 2011 Dec;30(12):1069-74. doi: 10.1097/INF.0b013e318234c886. PMID 22051859
- [Result] Williams PL, Seage GR 3rd, Van Dyke RB, Siberry GK, Griner R, Tassiopoulos K, Yildirim C, Read JS, Huo Y, Hazra R, Jacobson DL, Mofenson LM, Rich K; Pediatric HIV/AIDS Cohort Study. A trigger-based design for evaluating the safety of in utero antiretroviral exposure in uninfected children of human immunodeficiency virus-infected mothers. Am J Epidemiol. 2012 May 1;175(9):950-61. doi: 10.1093/aje/kwr401. Epub 2012 Apr 6. PMID 22491086
- [Result] Siberry GK, Williams PL, Mendez H, Seage GR 3rd, Jacobson DL, Hazra R, Rich KC, Griner R, Tassiopoulos K, Kacanek D, Mofenson LM, Miller T, DiMeglio LA, Watts DH; Pediatric HIV/AIDS Cohort Study (PHACS). Safety of tenofovir use during pregnancy: early growth outcomes in HIV-exposed uninfected infants. AIDS. 2012 Jun 1;26(9):1151-9. doi: 10.1097/QAD.0b013e328352d135. PMID 22382151
- [Result] Watts DH, Williams PL, Kacanek D, Griner R, Rich K, Hazra R, Mofenson LM, Mendez HA; Pediatric HIV/AIDS Cohort Study. Combination antiretroviral use and preterm birth. J Infect Dis. 2013 Feb 15;207(4):612-21. doi: 10.1093/infdis/jis728. Epub 2012 Nov 29. PMID 23204173
- [Result] Wilkinson JD, Williams PL, Leister E, Zeldow B, Shearer WT, Colan SD, Siberry GK, Dooley LB, Scott GB, Rich KC, Lipshultz SE; Pediatric HIVAIDS Cohort Study (PHACS). Cardiac biomarkers in HIV-exposed uninfected children. AIDS. 2013 Apr 24;27(7):1099-108. doi: 10.1097/QAD.0b013e32835cf21c. PMID 23211773
- [Result] Sirois PA, Huo Y, Williams PL, Malee K, Garvie PA, Kammerer B, Rich K, Van Dyke RB, Nozyce ML; Pediatric HIVAIDS Cohort Study. Safety of perinatal exposure to antiretroviral medications: developmental outcomes in infants. Pediatr Infect Dis J. 2013 Jun;32(6):648-55. doi: 10.1097/INF.0b013e318284129a. PMID 23340561
- [Result] Himes SK, Scheidweiler KB, Tassiopoulos K, Kacanek D, Hazra R, Rich K, Huestis MA; Pediatric HIV/AIDS Cohort Study. Development and validation of the first liquid chromatography-tandem mass spectrometry assay for simultaneous quantification of multiple antiretrovirals in meconium. Anal Chem. 2013 Feb 5;85(3):1896-904. doi: 10.1021/ac303188j. Epub 2013 Jan 14. PMID 23256731
- [Result] Rice ML, Zeldow B, Siberry GK, Purswani M, Malee K, Hoffman HJ, Frederick T, Buchanan A, Sirois PA, Allison SM, Williams PL; Pediatric HIVAIDS Cohort Study (PHACS). Evaluation of risk for late language emergence after in utero antiretroviral drug exposure in HIV-exposed uninfected infants. Pediatr Infect Dis J. 2013 Oct;32(10):e406-13. doi: 10.1097/INF.0b013e31829b80ee. PMID 24067563
- [Result] Malee KM, Mellins CA, Huo Y, Tassiopoulos K, Smith R, Sirois PA, Allison SM, Kacanek D, Kapetanovic S, Williams PL, Grant ML, Marullo D, Aidala AA; Pediatric HIVAIDS Cohort Study (PHACS). Prevalence, incidence, and persistence of psychiatric and substance use disorders among mothers living with HIV. J Acquir Immune Defic Syndr. 2014 Apr 15;65(5):526-34. doi: 10.1097/QAI.0000000000000070. PMID 24759063
- [Result] Nozyce ML, Huo Y, Williams PL, Kapetanovic S, Hazra R, Nichols S, Hunter S, Smith R, Seage GR 3rd, Sirois PA; Pediatric HIVAIDS Cohort Study. Safety of in utero and neonatal antiretroviral exposure: cognitive and academic outcomes in HIV-exposed, uninfected children 5-13 years of age. Pediatr Infect Dis J. 2014 Nov;33(11):1128-33. doi: 10.1097/INF.0000000000000410. PMID 25361407
- [Result] Williams PL, Crain MJ, Yildirim C, Hazra R, Van Dyke RB, Rich K, Read JS, Stuard E, Rathore M, Mendez HA, Watts DH; Pediatric HIV/AIDS Cohort Study. Congenital anomalies and in utero antiretroviral exposure in human immunodeficiency virus-exposed uninfected infants. JAMA Pediatr. 2015 Jan;169(1):48-55. doi: 10.1001/jamapediatrics.2014.1889. PMID 25383770
- [Result] Lipshultz SE, Williams PL, Zeldow B, Wilkinson JD, Rich KC, van Dyke RB, Seage GR 3rd, Dooley LB, Kaltman JR, Siberry GK, Mofenson LM, Shearer WT, Colan SD; Pediatric HIVAIDS Cohort Study (PHACS). Cardiac effects of in-utero exposure to antiretroviral therapy in HIV-uninfected children born to HIV-infected mothers. AIDS. 2015 Jan 2;29(1):91-100. doi: 10.1097/QAD.0000000000000499. PMID 25562493
- [Result] Rough K, Tassiopoulos K, Kacanek D, Griner R, Yogev R, Rich KC, Seage GR 3rd; Pediatric HIVAIDS Cohort Study. Dramatic decline in substance use by HIV-infected pregnant women in the United States from 1990 to 2012. AIDS. 2015 Jan 2;29(1):117-23. doi: 10.1097/QAD.0000000000000503. PMID 25562496
- [Result] Himes SK, Wu JW, Jacobson DL, Tassiopoulos K, Hazra R, Kacanek D, Van Dyke RB, Rich KC, Siberry GK, Huestis MA; Pediatric HIVAIDS Cohort Study (PHACS). Meconium Tenofovir Concentrations and Growth and Bone Outcomes in Prenatally Tenofovir Exposed HIV-Uninfected Children. Pediatr Infect Dis J. 2015 Aug;34(8):851-7. doi: 10.1097/INF.0000000000000747. PMID 25961889
- [Result] Himes SK, Huo Y, Siberry GK, Williams PL, Rice ML, Sirois PA, Frederick T, Hazra R, Huestis MA; Pediatric HIVAIDS Cohort Study. Meconium Atazanavir Concentrations and Early Language Outcomes in HIV-Exposed Uninfected Infants With Prenatal Atazanavir Exposure. J Acquir Immune Defic Syndr. 2015 Jun 1;69(2):178-86. doi: 10.1097/QAI.0000000000000558. PMID 26009830
- [Result] Himes SK, Tassiopoulos K, Yogev R, Huestis MA; Pediatric HIV/AIDS Cohort Study (PHACS). Antiretroviral Drugs in Meconium: Detection for Different Gestational Periods of Exposure. J Pediatr. 2015 Aug;167(2):305-11.e3. doi: 10.1016/j.jpeds.2015.04.062. Epub 2015 May 19. PMID 26001315
- [Result] Marsit CJ, Brummel SS, Kacanek D, Seage GR 3rd, Spector SA, Armstrong DA, Lester BM, Rich K; Pediatric HIV/AIDS Cohort Studies Network. Infant peripheral blood repetitive element hypomethylation associated with antiretroviral therapy in utero. Epigenetics. 2015;10(8):708-16. doi: 10.1080/15592294.2015.1060389. PMID 26067216
- [Result] Siberry GK, Jacobson DL, Kalkwarf HJ, Wu JW, DiMeglio LA, Yogev R, Knapp KM, Wheeler JJ, Butler L, Hazra R, Miller TL, Seage GR 3rd, Van Dyke RB, Barr E, Davtyan M, Mofenson LM, Rich KC; Pediatric HIV/AIDS Cohort Study. Lower Newborn Bone Mineral Content Associated With Maternal Use of Tenofovir Disoproxil Fumarate During Pregnancy. Clin Infect Dis. 2015 Sep 15;61(6):996-1003. doi: 10.1093/cid/civ437. Epub 2015 Jun 9. PMID 26060285
- [Result] Kirmse B, Yao TJ, Hofherr S, Kacanek D, Williams PL, Hobbs CV, Hazra R, Borkowsky W, Van Dyke RB, Summar M. Acylcarnitine Profiles in HIV-Exposed, Uninfected Neonates in the United States. AIDS Res Hum Retroviruses. 2016 Apr;32(4):339-48. doi: 10.1089/AID.2015.0112. Epub 2016 Jan 19. PMID 26548585
- [Result] Williams PL, Hazra R, Van Dyke RB, Yildirim C, Crain MJ, Seage GR 3rd, Civitello L, Ellis A, Butler L, Rich K; Pediatric HIV/AIDS Cohort Study. Antiretroviral exposure during pregnancy and adverse outcomes in HIV-exposed uninfected infants and children using a trigger-based design. AIDS. 2016 Jan 2;30(1):133-44. doi: 10.1097/QAD.0000000000000916. PMID 26731758
- [Result] Guerra V, Leister EC, Williams PL, Starc TJ, Lipshultz SE, Wilkinson JD, Van Dyke RB, Hazra R, Colan SD. Long-Term Effects of In Utero Antiretroviral Exposure: Systolic and Diastolic Function in HIV-Exposed Uninfected Youth. AIDS Res Hum Retroviruses. 2016 Jul;32(7):621-7. doi: 10.1089/AID.2015.0281. Epub 2016 May 9. PMID 26794032
- [Result] Caniglia EC, Patel K, Huo Y, Williams PL, Kapetanovic S, Rich KC, Sirois PA, Jacobson DL, Hernandez-Diaz S, Hernan MA, Seage GR 3rd; Pediatric HIVAIDS Cohort Study. Atazanavir exposure in utero and neurodevelopment in infants: a comparative safety study. AIDS. 2016 May 15;30(8):1267-78. doi: 10.1097/QAD.0000000000001052. PMID 26867136
- [Result] Van Dyke RB, Chadwick EG, Hazra R, Williams PL, Seage GR 3rd. The PHACS SMARTT Study: Assessment of the Safety of In Utero Exposure to Antiretroviral Drugs. Front Immunol. 2016 May 23;7:199. doi: 10.3389/fimmu.2016.00199. eCollection 2016. PMID 27242802
- [Result] Jacobson DL, Patel K, Williams PL, Geffner ME, Siberry GK, DiMeglio LA, Crain MJ, Mirza A, Chen JS, McFarland E, Kacanek D, Silio M, Rich K, Borkowsky W, Van Dyke RB, Miller TL; Pediatric HIVAIDS Cohort Study. Growth at 2 Years of Age in HIV-exposed Uninfected Children in the United States by Trimester of Maternal Antiretroviral Initiation. Pediatr Infect Dis J. 2017 Feb;36(2):189-197. doi: 10.1097/INF.0000000000001387. PMID 27798548
- [Result] Hermetet-Lindsay KD, Correia KF, Williams PL, Smith R, Malee KM, Mellins CA, Rutstein RM; Pediatric HIV/AIDS Cohort Study. Contributions of Disease Severity, Psychosocial Factors, and Cognition to Behavioral Functioning in US Youth Perinatally Exposed to HIV. AIDS Behav. 2017 Sep;21(9):2703-2715. doi: 10.1007/s10461-016-1508-5. PMID 27475941
- [Result] Tassiopoulos K, Huo Y, Braun J, Williams PL, Smith R, Aschengrau A, Nichols S, Hazra R, Meyer WA, Knapp K, Deygoo NS, Seage Iii GR. Blood lead levels and neurodevelopmental function in perinatally HIV-exposed, uninfected children in a US-based longitudinal cohort study. AIDS Res Hum Retroviruses. 2017 Sep;33(9):919-928. doi: 10.1089/AID.2016.0265. Epub 2017 Mar 21. PMID 28322573
- [Result] Jao J, Kacanek D, Williams PL, Geffner ME, Livingston EG, Sperling RS, Patel K, Bardeguez AD, Burchett SK, Chakhtoura N, Scott GB, Van Dyke RB, Abrams EJ; Pediatric HIV/AIDS Cohort Study and the International Maternal Pediatric Adolescent AIDS Clinical Trials P1025 Protocol; Pediatric HIV/AIDS Cohort Study and the International Maternal Pediatric Adolescent AIDS Clinical Trials P1025 Protocol. Birth Weight and Preterm Delivery Outcomes of Perinatally vs Nonperinatally Human Immunodeficiency Virus-Infected Pregnant Women in the United States: Results From the PHACS SMARTT Study and IMPAACT P1025 Protocol. Clin Infect Dis. 2017 Sep 15;65(6):982-989. doi: 10.1093/cid/cix488. PMID 28575201
- [Result] Rough K, Seage GR 3rd, Williams PL, Hernandez-Diaz S, Huo Y, Chadwick EG, Currier JS, Hoffman RM, Barr E, Shapiro DE, Patel K; PHACS and the IMPAACT P1025 Study Teams. Birth Outcomes for Pregnant Women with HIV Using Tenofovir-Emtricitabine. N Engl J Med. 2018 Apr 26;378(17):1593-1603. doi: 10.1056/NEJMoa1701666. PMID 29694825
- [Result] Goodenough CJ, Patel K, Van Dyke RB; Pediatric HIV/AIDS Cohort Study (PHACS). Is There a Higher Risk of Mother-to-child Transmission of HIV Among Pregnant Women With Perinatal HIV Infection? Pediatr Infect Dis J. 2018 Dec;37(12):1267-1270. doi: 10.1097/INF.0000000000002084. PMID 29742647
- [Result] Alperen J, Davidson J, Siminski S, Seage GR 3rd; Pediatric HIV/AIDS Cohort Study. Utility of the National Death Index in Identifying Deaths in a Clinic-Based, Multisite Cohort: The Experience of the Pediatric HIV/AIDS Cohort Study. J Acquir Immune Defic Syndr. 2018 Sep 1;79(1):e37-e39. doi: 10.1097/QAI.0000000000001763. No abstract available. PMID 29847477
- [Result] Jao J, Jacobson DL, Yu W, Borkowsky W, Geffner ME, McFarland EJ, Patel K, Williams PL, Miller T; Pediatric HIV/AIDS Cohort Study. A Comparison of Metabolic Outcomes Between Obese HIV-Exposed Uninfected Youth From the PHACS SMARTT Study and HIV-Unexposed Youth From the NHANES Study in the United States. J Acquir Immune Defic Syndr. 2019 Jul 1;81(3):319-327. doi: 10.1097/QAI.0000000000002018. PMID 30844997
- [Result] Margossian R, Williams PL, Yu W, Jacobson DL, Geffner ME, DiMeglio LA, Van Dyke RB, Spector SA, Schuster GU, Stephensen CB, Miller TL, Lipshultz SE; Pediatric HIV/AIDS Cohort Study (PHACS). Markers of Bone Mineral Metabolism and Cardiac Structure and Function in Perinatally HIV-Infected and HIV-Exposed but Uninfected Children and Adolescents. J Acquir Immune Defic Syndr. 2019 Jun 1;81(2):238-246. doi: 10.1097/QAI.0000000000002007. PMID 30865170
- [Result] Sudfeld CR, Jacobson DL, Rueda NM, Neri D, Mendez AJ, Butler L, Siminski S, Hendricks KM, Mellins CA, Duggan CP, Miller TL; Pediatric HIV/AIDS Cohort Study. Third Trimester Vitamin D Status Is Associated With Birth Outcomes and Linear Growth of HIV-Exposed Uninfected Infants in the United States. J Acquir Immune Defic Syndr. 2019 Jul 1;81(3):336-344. doi: 10.1097/QAI.0000000000002041. PMID 31021992
- [Result] Wang Y, Brummel SS, Beilstein-Wedel E, Dagnall CL, Hazra R, Kacanek D, Chadwick EG, Marsit CJ, Chanock SJ, Savage SA, Poirier MC, Machiela MJ, Engels EA; Pediatric HIV/AIDS Cohort Study. Association between zidovudine-containing antiretroviral therapy exposure in utero and leukocyte telomere length at birth. AIDS. 2019 Nov 1;33(13):2091-2096. doi: 10.1097/QAD.0000000000002317. PMID 31335808
- [Result] Purswani MU, Russell JS, Dietrich M, Malee K, Spector SA, Williams PL, Frederick T, Burchett S, Redmond S, Hoffman HJ, Torre P 3rd, Lee S, Rice ML, Yao TJ; Pediatric HIV/AIDS Cohort Study. Birth Prevalence of Congenital Cytomegalovirus Infection in HIV-Exposed Uninfected Children in the Era of Combination Antiretroviral Therapy. J Pediatr. 2020 Jan;216:82-87.e2. doi: 10.1016/j.jpeds.2019.09.025. Epub 2019 Oct 23. PMID 31668479
- [Result] Williams PL, Yildirim C, Chadwick EG, Van Dyke RB, Smith R, Correia KF, DiPerna A, Seage GR 3rd, Hazra R, Crowell CS; Surveillance Monitoring for ART Toxicities (SMARTT) study of the Pediatric HIV/AIDS Cohort Study. Association of maternal antiretroviral use with microcephaly in children who are HIV-exposed but uninfected (SMARTT): a prospective cohort study. Lancet HIV. 2020 Jan;7(1):e49-e58. doi: 10.1016/S2352-3018(19)30340-6. Epub 2019 Nov 15. PMID 31740351
- [Result] Powis KM, Huo Y, Williams PL, Kacanek D, Jao J, Patel K, Seage GR 3rd, Van Dyke RB, Chadwick EG; Pediatric HIV/AIDS Cohort Study (PHACS). Antiretroviral Prescribing Practices Among Pregnant Women Living With HIV in the United States, 2008-2017. JAMA Netw Open. 2019 Dec 2;2(12):e1917669. doi: 10.1001/jamanetworkopen.2019.17669. PMID 31851347
- [Result] Pintye J, Huo Y, Kacanek D, Zhang K, Kuncze K, Okochi H, Gandhi M. Extent of In Utero Transfer of Tenofovir From Mother to Fetus: A Paired Analysis of Hair Specimens Collected at Birth From a Cohort in the United States. J Infect Dis. 2021 Feb 24;223(4):638-644. doi: 10.1093/infdis/jiaa398. PMID 32620015
- [Result] Pintye J, Huo Y, Kacanek D, Zhang K, Kuncze K, Okochi H, Gandhi M; Pediatric HIV/AIDS Cohort Study (PHACS). Detectable HIV RNA in late pregnancy associated with low tenofovir hair levels at time of delivery among women living with HIV in the United States. AIDS. 2021 Feb 2;35(2):267-274. doi: 10.1097/QAD.0000000000002730. PMID 33055571
- [Result] O'Brien BE, Williams PL, Huo Y, Kacanek D, Chadwick EG, Powis KM, Correia K, Haddad LB, Yee LM, Chakhtoura N, Dola C, Van Dyke RB; Pediatric HIV/AIDS Cohort Study (PHACS). Repeat Pregnancies Among US Women Living With HIV in the SMARTT Study: Temporal Changes in HIV Disease Status and Predictors of Preterm Birth. J Acquir Immune Defic Syndr. 2020 Nov 1;85(3):346-354. doi: 10.1097/QAI.0000000000002445. PMID 32701825
- [Result] Torre P Rd, Zeldow B, Yao TJ, Hoffman HJ, Siberry GK, Purswani MU, Frederick T, Spector SA, Williams PL. Newborn Hearing Screenings in Human Immunodeficiency Virus-Exposed Uninfected Infants. J AIDS Immune Res. 2016;1(1):102. Epub 2016 Sep 5. PMID 28459118
- [Result] Rice ML, Russell JS, Frederick T, Purswani M, Williams PL, Siberry GK, Redmond SM, Hoffman HJ, Yao TJ; Pediatric HIV/AIDS Cohort Study (PHACS). Risk for Speech and Language Impairments in Preschool Age HIV-exposed Uninfected Children With In Utero Combination Antiretroviral Exposure. Pediatr Infect Dis J. 2018 Jul;37(7):678-685. doi: 10.1097/INF.0000000000001875. PMID 29278615
- [Result] Miller TL, Jacobson DL, Somarriba G, Neri D, Kurtz-Vraney J, Graham P, Gillman MW, Landy DC, Siminski S, Butler L, Rich KC, Hendricks K, Ludwig DA; Pediatric HIV/AIDS Cohort Study. A multicenter study of diet quality on birth weight and gestational age in infants of HIV-infected women. Matern Child Nutr. 2017 Oct;13(4):e12378. doi: 10.1111/mcn.12378. Epub 2016 Nov 8. PMID 27863014
- [Result] Williams PL, Huo Y, Rutstein R, Hazra R, Rough K, Van Dyke RB, Chadwick EG. Trends in Neonatal Prophylaxis and Predictors of Combination Antiretroviral Prophylaxis in US Infants from 1990 to 2015. AIDS Patient Care STDS. 2018 Feb;32(2):48-57. doi: 10.1089/apc.2017.0295. PMID 30346801
- [Result] Jao J, Kacanek D, Yu W, Williams PL, Patel K, Burchett S, Scott G, Abrams EJ, Sperling RS, Van Dyke RB, Smith R, Malee K; Pediatric HIV/AIDS Cohort Study. Neurodevelopment of HIV-Exposed Uninfected Infants Born to Women With Perinatally Acquired HIV in the United States. J Acquir Immune Defic Syndr. 2020 Jun 1;84(2):213-219. doi: 10.1097/QAI.0000000000002318. PMID 32032301
- [Result] Crowell CS, Williams PL, Yildirim C, Van Dyke RB, Smith R, Chadwick EG, Seage GR 3rd, Diperna A, Hazra R; Pediatric HIV/AIDS Cohort Study. Safety of in-utero antiretroviral exposure: neurologic outcomes in children who are HIV-exposed but uninfected. AIDS. 2020 Jul 15;34(9):1377-1387. doi: 10.1097/QAD.0000000000002550. PMID 32310900
- [Result] Labuda SM, Huo Y, Kacanek D, Patel K, Huybrechts K, Jao J, Smith C, Hernandez-Diaz S, Scott G, Burchett S, Kakkar F, Chadwick EG, Van Dyke RB; Pediatric HIV/AIDS Cohort Study. Rates of Hospitalization and Infection-Related Hospitalization Among Human Immunodeficiency Virus (HIV)-Exposed Uninfected Children Compared to HIV-Unexposed Uninfected Children in the United States, 2007-2016. Clin Infect Dis. 2020 Jul 11;71(2):332-339. doi: 10.1093/cid/ciz820. PMID 31504291
- [Result] Lin SH, Wang Y, Hartley SW, Karyadi DM, Lee OW, Zhu B, Zhou W, Brown DW, Beilstein-Wedel E, Hazra R, Kacanek D, Chadwick EG, Marsit CJ, Poirier MC, Brummel SS, Chanock SJ, Engels EA, Machiela MJ; Pediatric HIV/AIDS Cohort Study. In-utero exposure to zidovudine-containing antiretroviral therapy and clonal hematopoiesis in HIV-exposed uninfected newborns. AIDS. 2021 Aug 1;35(10):1525-1535. doi: 10.1097/QAD.0000000000002894. PMID 33756513
- [Result] Jacobson DL, Neri D, Gaskins A, Yee L, Mendez AJ, Hendricks K, Siminski S, Zash R, Hyzy L, Jao J; Pediatric HIV/AIDS Cohort Study. Maternal anemia and preterm birth among women living with HIV in the United States. Am J Clin Nutr. 2021 Jun 1;113(6):1402-1410. doi: 10.1093/ajcn/nqaa441. PMID 35104854
- [Result] Smith C, Huo Y, Patel K, Fetters K, Hegemann S, Burchett S, Van Dyke R, Weinberg A. Immunologic and Virologic Factors Associated With Hospitalization in Human Immunodeficiency Virus-Exposed, Uninfected Infants in the United States. Clin Infect Dis. 2021 Sep 15;73(6):1089-1096. doi: 10.1093/cid/ciab272. PMID 34157096
- [Result] Yee LM, Kacanek D, Brightwell C, Haddad LB, Jao J, Powis KM, Yao TJ, Barr E, Broadwell C, Siminski S, Seage GR 3rd, Chadwick EG; Pediatric HIV/AIDS Cohort Study. Marijuana, Opioid, and Alcohol Use Among Pregnant and Postpartum Individuals Living With HIV in the US. JAMA Netw Open. 2021 Dec 1;4(12):e2137162. doi: 10.1001/jamanetworkopen.2021.37162. PMID 34860242
- [Result] Yu W, Jacobson DL, Williams PL, Patel K, Geffner ME, Van Dyke RB, Kacanek D, DiMeglio LA, Jao J; Pediatric HIV/AIDS Cohort Study (PHACS). Growth patterns of uninfected children born to women living with perinatally versus nonperinatally acquired HIV. AIDS. 2022 Mar 15;36(4):593-603. doi: 10.1097/QAD.0000000000003136. PMID 34860195
- [Result] Young MR, Broadwell C, Kacanek D, Chadwick EG, Jao J, Moscicki AB, Powis K, Tassiopoulos K, Yee LM, Haddad LB; Pediatric HIV/AIDS Cohort Study. Sexually Transmitted Infections in Pregnant People With Human Immunodeficiency Virus: Temporal Trends, Demographic Correlates, and Association With Preterm Birth. Clin Infect Dis. 2022 Dec 19;75(12):2211-2218. doi: 10.1093/cid/ciac321. PMID 35486952
- [Result] Yee LM, Jacobson DL, Haddad LB, Jao J, Powis KM, Kacanek D, Zash R, DiPerna A, Chadwick EG; Pediatric HIV/AIDS Cohort Study. Evaluating the association of antiretroviral therapy and immune status with hypertensive disorders of pregnancy among people with HIV. AIDS. 2023 Sep 1;37(11):1715-1723. doi: 10.1097/QAD.0000000000003607. Epub 2023 May 23. PMID 37260289
- [Result] Jao J, Kacanek D, Broadwell C, Jacobson DL, Chadwick EG, Williams PL, Powis KM, Haddad LB, Yee L; Pediatric HIV/AIDS Cohort Study. Gestational weight gain in persons with HIV in the United States. AIDS. 2023 May 1;37(6):883-893. doi: 10.1097/QAD.0000000000003454. Epub 2022 Dec 2. PMID 36729961
- [Result] Shiau S, Jacobson DL, Huo Y, Kacanek D, Yee LM, Williams DB, Haddad LB, Serghides L, Powis K, Sperling RS, Williams PL, Jao J; Pediatric HIV/AIDS Cohort Study. Unique Profile of Inflammation and Immune Activation in Pregnant People With HIV in the United States. J Infect Dis. 2023 Mar 1;227(5):720-730. doi: 10.1093/infdis/jiac501. PMID 36592383
- [Result] Yao TJ, Malee K, Zhang J, Smith R, Redmond S, Rice ML, Frederick T, Torre P, Mellins CA, Hoffman HJ, Williams PL. In Utero Antiretroviral Exposure and Risk of Neurodevelopmental Problems in HIV-Exposed Uninfected 5-Year-Old Children. AIDS Patient Care STDS. 2023 Mar;37(3):119-130. doi: 10.1089/apc.2022.0189. Epub 2023 Feb 24. PMID 36827595
- [Result] Davtyan M, Kacanek D, Lee J, Berman C, Chadwick EG, Smith R, Salomon L, Frederick T; Pediatric HIV/AIDS Cohort Study. The role of internalised HIV stigma in disclosure of maternal HIV serostatus to children perinatally HIV-exposed but uninfected: a prospective study in the United States. J Int AIDS Soc. 2023 Oct;26 Suppl 4(Suppl 4):e26167. doi: 10.1002/jia2.26167. PMID 37909234
- [Result] Davtyan M, Kacanek D, Lee J, Berman C, Chadwick EG, Smith R, Salomon L, Frederick T; Pediatric HIV/AIDS Cohort Study. Factors associated with internalized HIV-related stigma among biological mothers living with HIV enrolled in a US cohort study. AIDS Care. 2024 Feb;36(2):220-226. doi: 10.1080/09540121.2023.2263680. Epub 2024 Jan 30. PMID 37757482
- [Result] Fisher SA, Jao JK, Yee LM, Serghides L, Chadwick EG, Jacobson DL. Association of Fatty Acid Signatures with HIV Viremia in Pregnancy. AIDS Res Hum Retroviruses. 2024 Apr;40(4):257-267. doi: 10.1089/AID.2023.0040. Epub 2023 Oct 30. PMID 37772708
- [Result] Berhie S, Kacanek D, Lee J, Jao J, Powis K, Salomon L, Siddiqui D, Yee LM; Pediatric HIV/AIDS Cohort Study. Routine Vaccination During Pregnancy Among People Living With HIV in the United States. JAMA Netw Open. 2024 May 1;7(5):e249531. doi: 10.1001/jamanetworkopen.2024.9531. PMID 38696165
- [Result] Fung K, Hernandez-Diaz S, Zash R, Chadwick EG, Van Dyke RB, Broadwell C, Jao J, Powis K, Yee LM, Williams PL; Pediatrics HIV/AIDS Cohort Study (PHACS). First-trimester exposure to newer antiretroviral agents and congenital anomalies in a US cohort. AIDS. 2024 Sep 1;38(11):1686-1695. doi: 10.1097/QAD.0000000000003955. Epub 2024 Jun 11. PMID 38864586
- [Result] Purswani MU, Jacobson DL, DiMeglio LA, Yao TJ, Kopp JB, Van Dyke RB, Yu W, Siberry GK; Pediatric HIV/AIDS Cohort Study (PHACS). Phosphaturia in HIV-Exposed Uninfected Neonates Associated with Maternal Use of Tenofovir Disoproxil Fumarate in Late Pregnancy. J Pediatric Infect Dis Soc. 2024 Aug 24;13(8):396-405. doi: 10.1093/jpids/piae054. PMID 38820092
- [Result] Gojanovich GS, Marsit CJ, Kacanek D, Russell J, Hudson G, Van Dyke RB, Naini AB, Gerschenson M; Pediatric HIV/AIDS Cohort Study. Relationships of mitochondrial DNA mutations and select clinical diagnoses in perinatally HIV- and ART-exposed uninfected children. Mitochondrion. 2024 Nov;79:101949. doi: 10.1016/j.mito.2024.101949. Epub 2024 Aug 30. PMID 39218053
- [Result] Olivero R, Williams PL, Sawyer G, Yee LM, Patel K, Hernandez-Diaz S, Powis K, Paul M, Chadwick EG; Pediatric HIV/AIDS Cohort Study and the HOPE study. Birth outcomes following bictegravir exposure during pregnancy. AIDS. 2025 Mar 15;39(4):381-386. doi: 10.1097/QAD.0000000000004041. Epub 2024 Oct 14. PMID 39411892
- See also: Pediatric HIV/AIDS Cohort Study — https://www.phacsstudy.org